CLINICAL TRIAL: NCT01218295
Title: Efficacy of Inspiratory Muscle Training by Means of Spirotiger® in COPD Patients.
Brief Title: Inspiratory Muscle Training With Normocapnic Hyperpnea in Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Annalisa Cogo, University of Ferrara
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMTCOPD2
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-10

CONDITIONS: COPD
Keywords: COPD; inspiratory muscles training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Respiratory muscle training (Experimental): Patients assigned to this arm train the respiratory muscles by means of normocapnic hyperpnea.
  Interventions: Device: Spirotiger®

INTERVENTIONS:
Device: Spirotiger® — training session :10 minutes twice a day X 4 weeks
  Other Names: Pulmonary rehabilitation

SUMMARY:
Many studies suggest that inspiratory muscles training by means of normocapnic hyperpnea improves exercise tolerance in healthy subjects. No information is available about the use of this training in COPD patients even if other methods (such as threshold loading and resistive loading) have been shown to be effective in terms of Inspiratory Muscle Function, Health-Related Quality of Life and Exercise Tolerance.

This study is designed to evaluate the effects of normocapnic hyperventilation by means of Spirotiger®, an instrument training the respiratory muscles, avoiding hypocapnia (using the methodology of isocapnic hyperpnoea)in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients. All patients are at stable state, free from an exacerbation from at least 3 months.

Exclusion Criteria:

* COPD patients with a recent history of cardiovascular disease, neurologic disease and other diseases that would interfere with the training.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Exercise Capacity | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Annalisa Cogo, MD, Principal Investigator — Università di Ferrara
Locations (1):
- Pulmonary Respiratory Unit- University Hospital, Ferrara, Ferrara, Italy